CLINICAL TRIAL: NCT06600438
Title: Slowing Parkinson's Early Through Exercise Dosage - United Kingdom
Brief Title: Slowing Parkinson's Early Through Exercise Dosage-United Kingdom
Acronym: Slow-SPEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 362207
Record Dates: First submitted 2024-07-22; First posted 2024-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hyposmia; Anosmia
Keywords: Parkinson's Disease; Parkinson Disease; Anosmia; Hyposmia; Smell loss; Exercise; Prevention
MeSH Terms: conditions — Anosmia; Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100% exercise increase (Experimental): Arm: Full-Dose Exercise Group Participants in this arm will be asked to increase their average daily step count by 100% compared with baseline. Using a Fitbit smartwatch and the Slow-SPEED smartphone app, they will receive personalised step goals, real-time feedback, and gamified challenges to encourage gradual and sustained increases in physical activity. The programme is delivered remotely and unsupervised over 18 months, with progress monitored continuously through the wearable device.
  Interventions: Other: Slow-SPEED app
- 10% exercise increase (Active Comparator): Arm: Low-Dose Control Group Participants in this arm will be asked to increase their average daily step count by 10% compared with baseline. Like the intervention group, they will use a Fitbit smartwatch and the Slow-SPEED smartphone app, receiving similar gamified feedback and motivational tools. The lower step target provides an active control condition while maintaining blinding. The programme is delivered remotely and unsupervised over 18 months, with continuous monitoring via the wearable device.
  Interventions: Other: Slow-SPEED app

INTERVENTIONS:
Other: Slow-SPEED app — Gamified motivational smartphone app

SUMMARY:
Parkinson's disease (PD) is the fastest growing neurological condition worldwide and currently has no treatment that slows or prevents it. Research shows that regular exercise may help protect the brain and delay symptoms. This study will test whether a long-term, home-based exercise programme can help people who are at increased risk of Parkinson's because they have a reduced sense of smell (called "hyposmia"). Hyposmia is a common early sign that can appear years before the movement symptoms of Parkinson's.

The study, called Slow-SPEED UK, will recruit 110 adults aged 40 and over who have hyposmia and are currently not very active (walking less than 7,000 steps a day). Participants will first complete a four-week baseline period to confirm eligibility, then be randomly assigned (like flipping a coin) to one of two groups:

Full-dose exercise group - encouraged to gradually double their daily step count using a fitness tracker and smartphone app.

Low-dose control group - encouraged to increase daily steps by 10% using the same tools.

Both groups will use the study's fitness tracker and app, which provides goals, feedback, and motivation through gamification. The programme lasts 18 months, with assessments at the start, mid-point (9 months), and end (18 months). Some participants may also give optional blood or skin samples to help researchers explore biological changes linked to early Parkinson's.

The main question this study will answer is whether a remote, app-based programme can successfully increase daily step counts in people with hyposmia. Researchers will also look at whether exercise affects other outcomes such as exercise intensity, mood, sleep, smell, movement, quality of life, and early biological markers of Parkinson's.

The study is designed as a feasibility trial. This means its main goal is to test whether the programme is practical, acceptable, and safe for participants. Results will inform larger future studies that could test whether structured exercise can delay or prevent Parkinson's disease in at-risk groups. Because exercise is already known to have many health benefits, all participants are expected to gain from taking part, regardless of whether they eventually develop Parkinson's.

DETAILED DESCRIPTION:
Background and Rationale:

Parkinson's disease (PD) is the fastest growing neurological disorder worldwide, and there are still no treatments proven to slow or prevent it. By the time PD is diagnosed, most dopamine-producing neurons in the brain are already lost. This highlights the importance of testing preventive strategies during the prodromal (early) stage, before movement symptoms appear.

One of the most common prodromal features is hyposmia (reduced sense of smell), which is present in up to 90% of people who later develop PD. Individuals with hyposmia have nearly a fourfold increased risk of developing PD, making this group an ideal target for prevention-focused research.

Evidence from laboratory and clinical studies suggests that exercise may have protective effects on the brain by promoting neuroplasticity, reducing inflammation, and improving cellular health. Exercise is already known to improve mobility, mood, sleep, and quality of life in people with PD. Observational studies also show that more active individuals are less likely to develop PD. However, structured, long-term exercise trials have not yet been conducted in hyposmic individuals at risk of PD.

Study Objectives:

The primary objective is to test the feasibility of a remote, app-based exercise programme to increase daily step counts in adults with hyposmia. Secondary objectives include examining exercise intensity, digital fitness and gait markers, smell, sleep, mood, quality of life, and optional biomarkers of PD risk. This feasibility trial will inform the design of future large-scale studies.

Study Design:

Slow-SPEED UK is a two-arm, double-blind randomised controlled trial that will recruit 110 participants aged 40 years and older with confirmed hyposmia.

All participants complete a 4-week baseline period with a Fitbit device to confirm activity levels.

Eligible participants (average <7,000 steps/day) will be randomised 1:1 to:

Full-dose group: goal to double daily steps (100% increase).

Low-dose control group: goal to increase steps by 10%.

Both groups receive the Slow-SPEED smartphone app and Fitbit, which provide gamified feedback, challenges, and motivation.

Follow-up assessments occur at baseline (in-person), 9 months (remote), and 18 months (in-person).

A subgroup will also provide blood and skin samples for exploratory biomarker studies.

The primary outcome is change in average daily step count from baseline to 18 months. Secondary measures include exercise intensity, free-living gait metrics, olfactory testing, patient-reported outcomes, and optional biomarkers.

Duration:

Each participant is enrolled for approximately 19 months (including the 4-week baseline and 18-month intervention). Recruitment is expected to take 5 months, for a total study length of about 2 years.

Risks and Benefits:

The risks are low and mainly relate to normal physical activity, such as mild muscle soreness or fatigue. Safety screening and eligibility criteria minimise risk. Unlike drug-based trials, there are no medication side effects.

The benefits are broad. Participants may gain improvements in mobility, sleep, and wellbeing regardless of PD risk. At a scientific level, the study will provide key information on whether long-term, remote exercise programmes are practical, acceptable, and safe for people with hyposmia, and whether they show early signals of benefit.

International Collaboration:

Slow-SPEED UK is part of Slow-SPEED International, a coordinated programme with parallel trials in the Netherlands (focusing on people with REM sleep behaviour disorder) and the USA (focusing on people with genetic PD risk variants such as LRRK2 or GBA1). By aligning protocols and outcome measures, the programme will enable pooled analyses across different prodromal groups. Together, these studies will build the evidence base for exercise as a low-cost, scalable strategy to delay or prevent Parkinson's disease worldwide.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 40 years
* Objective hyposmia, defined as scoring below the 15th percentile (adjusted for age/sex) on UPSIT
* Ability and willingness to provide written informed consent
* Proficiency in written and spoken English sufficient to complete study procedures.
* Willingness and ability to attend baseline (in-person), 9-month (remote), and 18-month (in-person) assessments.
* Access to telephone or internet for interim communication. Specifically, in possession of a suitable smartphone (screen size minimum 4.6 inch; Android version 9 or iOS version 15 or newer).
* Physical activity threshold: During the 4-week eligibility run-in, the mean daily step count must be <7,000 steps/day, calculated over ≥21 valid days (a valid day = ≥10 hours wear time or ≥1,000 steps). If recruitment after the first 2 months is <60-70% of target, and subject to TSC/Sponsor approval and REC amendment, eligibility may be broadened to <10,000 steps/day (i.e. participants averaging 7,000-9,999 steps/day become eligible).

Exclusion criteria

* Clinical diagnosis of PD, dementia, or other neurodegenerative conditions
* Severe or unstable medical or psychiatric illness likely to impair participation
* Use of agents known to alter olfaction (e.g. intranasal zinc, chronic corticosteroids)
* Current enrolment in an interventional study within the past 3 months (standard research retention guidance).
* Inability to complete study procedures in English, per investigator assessment
* Unable to give consent
* Participants not living independently in the community. Participants in nursing homes, hospitalised persons on in a non-institutionalised setting are excluded.
* Subject's personal smartphone is Fitbit-incompatible i.e. Huawei P8 Lite; Huawei P9 Lite; Xiaomi Mi 6; Huawei P20 Lite
* Activity level above threshold during eligibility run-in: mean daily step count ≥7,000 steps/day (or ≥10,000 steps/day if the broadened threshold is activated).

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in average daily step count | Baseline (weeks 0-4) to 18 months (weeks 75-78)
  Change in mean daily step count from baseline (weeks 0-4) to the final four weeks of the 18-month intervention (weeks 75-78), measured continuously using a Fitbit smartwatch. Step count is an objective, scalable measure of physical activity, validated in Parkinson's disease (PD) cohorts.

SECONDARY OUTCOMES:
Change in moderate-to-vigorous physical activity (MVPA) | Baseline, 9 months, and 18 months
  Change in minutes per week spent in MVPA (≥64% of age-predicted maximum heart rate), measured continuously by Fitbit smartwatch.
Digital markers of physical fitness | Continuous (Fitbit) and daily (phone PPG for VO₂max)
  Wearable-derived fitness metrics including resting heart rate, heart rate variability, gait composites, and VO₂max estimates. These reflect changes in free-living activity and cardiorespiratory fitness.
Motor outcomes | Baseline, every 6 weeks (Roche app), and 18 months
  Change in motor symptoms measured by Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS Part III), Functional Gait Assessment (FGA), Mini-BESTest, and Roche Mobile App V2 (digital motor assessments such as tapping, gait, tremor).
Non-motor and autonomic outcomes | Baseline, 9 months, and 18 months
  Composite assessments of autonomic symptoms (SCOPA-AUT), orthostatic hypotension, mood, sleep, and cognition (MoCA). Collected through in-person visits and questionnaires.
Change in health-related quality of life as measured by EQ-5D-5L and PDQ-39 scores between baseline and 18 months | Baseline and 18 months
  Patient-reported outcomes using validated tools including EQ-5D-5L and PDQ-39, administered digitally or in clinic.
Patient engagement and feasibility | Continuous throughout intervention
  Usability of the Slow-SPEED app, adherence to Fitbit wear time, completion of digital assessments, and retention in the study.
Laboratory biomarkers | Baseline and 18 months (subgroup only). Optional for participants
  Plasma and serum assays of α-synuclein species, neurofilament light (NfL), and inflammatory markers. Samples processed in duplicate with internal QC and false discovery rate correction.
Digital engagement metrics | Continuous across intervention
  Patterns of Fitbit wear time, app usage, weekly goal adherence, and interactions with motivational features of the Slow-SPEED app.
Prodromal Load Score (PLS) | Baseline, 9 months, and 18 months
  Composite index of cumulative prodromal burden (olfaction, sleep, autonomic features, mood, subtle motor changes). Derived and validated across international cohorts (PREDICT-PD, OPDC, Rotterdam, NAPS).
NeuroClues | Baseline (weeks 0-4) to 18 months (weeks 75-78)
  A non-invasive assessment tool. The NeuroClues system uses high-frequency binocular eye-tracking to capture objective measures of oculomotor control. The protocol involves a short calibration followed by a standardised battery of tasks (prosaccades, antisaccades, fixation and pursuit), with total testing time approximately 10-15 minutes. The tool automatically records and processes key endpoints including prosaccade latency (ms), antisaccade latency (ms), antisaccade error rate (%), fixation stability measures and saccadic intrusions.

CONTACTS AND LOCATIONS:
Overall Officials: Alastair J Noyce, BMedSci, MBBS, MSc, MRCP, PhD, Principal Investigator — Centre for Preventive Neurology, Queen Mary University of London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Slow-SPEED-UK participants will be identified via PREDICT-PD. — https://www.predictpd.com/
- See also: Slow-SPEED UK participants will be identified via the The Smell & Taste Clinic ENT Department James Paget University Hospital NHS Foundation Trust via collaborator: Professor Carl Philpott, Gorleston, Great Yarmouth Norfolk, NR31 6LA — https://www.jpaget.nhs.uk/departments/ear-nose-and-throat/